CLINICAL TRIAL: NCT02817503
Title: Effects of Intensive Antihypertensive Therapies on the Risk of Stroke in Hypertensive Adults: A Prospective Randomized Open-Label Blinded-Endpoint Trial, a Feasibility Study
Brief Title: Feasibility Study of the Intensive Systolic Blood Pressure Control
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Collaborators: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Xiaoshu Cheng, Professor, Second Affiliated Hospital of Nanchang University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20151BDH80038
Record Dates: First submitted 2016-06-18; First posted 2016-06-29 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Hypertension; Hyperhomocysteinemia
Keywords: hypertension; BP titration; intensive blood pressure control; primary prevention; China; H-type Hypertension
MeSH Terms: conditions — Hypertension; Hyperhomocysteinemia | interventions — Hydrochlorothiazide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard BP control (Experimental): SBP within 140 - <150 mmHg. For all participants, enalapril-folic acid will be used as an initial therapy. Other drugs, including CCB (amlodipine preferred), diuretics (hydrochlorothiazide preferred), and β-blockers, are allowed, in order to achieve the SBP target. For those who can't tolerate enalapril-folic acid well, other types of antihypertensive agents may be used as alternative choices.
  If the target BP level is not achieved during the Titration or Follow-up periods, adjustment of drug type and dosage will be carried out according to procedures defined in the protocol.
  Interventions: Drug: Standard BP control
- Moderate BP control (Active Comparator): SBP within 130 - <140 mmHg. For all participants, enalapril-folic acid will be used as an initial therapy. Other drugs, including CCB (amlodipine preferred), diuretics (hydrochlorothiazide preferred), and β-blockers, are allowed, in order to achieve the SBP target. For those who can't tolerate enalapril-folic acid well, other types of antihypertensive agents may be used as alternative choices.
  If the target BP level is not achieved during the Titration or Follow-up periods, adjustment of drug type and dosage will be carried out according to procedures defined in the protocol.
  Interventions: Drug: Moderate BP control
- Intensive BP control (Active Comparator): SBP <130 mmHg. For all participants, enalapril-folic acid will be used as an initial therapy. Other drugs, including CCB (amlodipine preferred), diuretics (hydrochlorothiazide preferred), and β-blockers, are allowed, in order to achieve the SBP target. For those who can't tolerate enalapril-folic acid well, other types of antihypertensive agents may be used as alternative choices.
  If the target BP level is not achieved during the Titration or Follow-up periods, adjustment of drug type and dosage will be carried out according to procedures defined in the protocol.
  Interventions: Drug: Intensive BP control

INTERVENTIONS:
Drug: Standard BP control — Enalapril-folic acid will be used as an initial therapy. Other drugs, including CCB (amlodipine preferred), diuretics (hydrochlorothiazide preferred), and β-blockers, are allowed, in order to achieve the SBP target.
  Other Names: Enalapril-folic acid,amlodipine,hydrochlorothiazide
  Arms: Standard BP control
Drug: Moderate BP control — Enalapril-folic acid will be used as an initial therapy. Other drugs, including CCB (amlodipine preferred), diuretics (hydrochlorothiazide preferred), and β-blockers, are allowed, in order to achieve the SBP target.
  Other Names: Enalapril-folic acid,amlodipine,hydrochlorothiazide
  Arms: Moderate BP control
Drug: Intensive BP control — Enalapril-folic acid will be used as an initial therapy. Other drugs, including CCB (amlodipine preferred), diuretics (hydrochlorothiazide preferred), and β-blockers, are allowed, in order to achieve the SBP target.
  Other Names: Enalapril-folic acid,amlodipine,hydrochlorothiazide
  Arms: Intensive BP control

SUMMARY:
The purpose of the current feasibility study is to test whether the blood pressure level of the study patients can be effectively and safely managed according to the intensive antihypertensive treatment protocol. Furthermore, the study will also examine the effect of intensive antihypertensive treatment on the intermediate cardiovascular diseases outcomes, including CIMT, carotid plaques, PWV ABI, and kidney function, etc.

DETAILED DESCRIPTION:
The China Stroke Primary Prevention Trial (CSPPT, NCT00794885) found that among hypertensive adults in China without a history of stroke or myocardial infarction, the combined use of enalapril and folic acid, compared with enalapril alone, significantly reduced the risk of first stroke. The mean systolic blood pressures were highly comparable between the two groups over the course of the trial (139.7mmHg and 139.8mmHg, respectively, in the enalapril-folic acid and the enalapril group). In the further analysis, lower systolic blood pressures seemed to be associated with greater reduction in cardiovascular outcomes in both of the treatment groups.

However, due to inconsistencies in the results of the ACCORD and SPRINT trials, the appropriate targets for systolic blood pressure in effectively reducing cardiovascular events among hypertensive patients remain uncertain.

The proposed trial aims to test the hypothesis that among hypertensive patients aged 60 years or older, a lower systolic blood pressure goal will lead to greater reduction in stroke incidence.

The current feasibility study aims to test whether the blood pressure level of the study patients can be effectively and safely managed according to the intensive antihypertensive treatment protocol. Furthermore, the study will also examine the effect of intensive antihypertensive treatment on the intermediate cardiovascular diseases outcomes, including CIMT, carotid plaques, PWV ABI, and kidney function, etc.

The current feasibility study will enroll approximately 100 patients with H-type hypertension (hypertensive patients with hyperhomocysteinemia) aged 60 years or older, and without a history of major cardiovascular diseases.

Eligible patients will randomly assigned to one of three different systolic blood pressure (SBP) target groups (Group A, SBP: 140 - <150 mmHg; Group B, SBP: 130 - < 140 mmHg; and Group C, SBP < 130 mmHg).

ELIGIBILITY:
Inclusion criteria:

* Hypertensive patients aged 60 years or older.
* SBP>= 150 mmHg but <180 mmHg, if currently (within the previous two weeks) not regularly treated with antihypertensive drugs.
* If currently (at least 10 days on medications within the previous two weeks) regularly treated with antihypertensive drugs, blood pressure must meet the following criteria:

SBP >= 140 mmHg but <170 mmHg, if regularly (no less than 10 days) taking 1 type of antihypertensive medication within the previous two weeks; SBP >= 130 mmHg but <160 mmHg, if regularly (no less than 10 days) taking 2 types of antihypertensive medications within the previous two weeks; SBP >= 130 mmHg but <150 mmHg, if regularly (no less than 10 days) taking 3 types of antihypertensive medication within the previous two weeks.

For patients taking a fixed-dose-combination (FDC), this treatment will be considered as two types of drugs if the dose of each component of the FDC is equal to higher than the routine therapeutic dose.

* Blood homocysteine (Hcy)≥ 10μmol/L, or the patient is taking enalapril-folic acid;
* Subject has read and signed a written, informed consent form.

Exclusion Criteria:

* History of physician diagnosed stroke, myocardial infarction, heart failure, revascularization, or malignancy;
* Clearly diagnosed secondary hypertension;
* Undergoing regular renal dialysis or has been diagnosed with end-stage kidney disease;
* Congenital or acquired organic heart disease;
* Severe somatic disease preventing the participant from completing the trial, or based on the discretion of the investigators, the patient is incapable of participating;
* Contraindicated or intolerable to ACEIs (including enalapril-folic acid) or a history of severe adverse effects to ACEIs;
* Individuals with abnormal laboratory test results and/or clinical manifestations rendering them unsuitable to participate as judged by the investigators;
* Any factor likely to limit adherence to interventions or jeopardize data collection, for example: dementia, severe mental disorders impeding expression or communication abilities, an inability to adhere the follow-up plan, plans to move in the near future, or, a history of unreliability in following a medication regimen or in keeping appointments;
* Living with a family member (a spouse, for example) who has already participated in the study;
* Unwilling to participate, unwilling or unable to change current therapeutic regimen;
* Currently (or within one month) participating in another new drug trial.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Achieved mean blood pressure levels in each of the treatment groups | 6 months BP titration treatment period

SECONDARY OUTCOMES:
Carotid intima-media thickness (CIMT), Carotid plaques | 6 months BP titration treatment period
Carotid-femoral pulse wave velocity, Brachial-ankle pulse wave velocity | 6 months BP titration treatment period
Ankle brachial index | 6 months BP titration treatment period
Urinary albumin-creatinine ratio | 6 months BP titration treatment period

OTHER OUTCOMES:
Events related to the intensive blood pressure control, Hypotension, Syncope, Bradycardia or Arrhythmia, Hyperkalemia, Renal Failure | 6 months BP titration treatment period
First Occurrence of a Major Cardiovascular Event (MCE); Specifically Nonfatal Heart Attack, Nonfatal Stroke, or Cardiovascular Death hospitalization; Hospitalization | during the Randomization and Titration Treatment period
  6 months BP titration treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoshu Cheng, MD, Principal Investigator — Second Affiliated Hospital of Nanchang University
Locations (1):
- the People's Hospital of Rongcheng, Yatou, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huo Y, Li J, Qin X, Huang Y, Wang X, Gottesman RF, Tang G, Wang B, Chen D, He M, Fu J, Cai Y, Shi X, Zhang Y, Cui Y, Sun N, Li X, Cheng X, Wang J, Yang X, Yang T, Xiao C, Zhao G, Dong Q, Zhu D, Wang X, Ge J, Zhao L, Hu D, Liu L, Hou FF; CSPPT Investigators. Efficacy of folic acid therapy in primary prevention of stroke among adults with hypertension in China: the CSPPT randomized clinical trial. JAMA. 2015 Apr 7;313(13):1325-35. doi: 10.1001/jama.2015.2274. PMID 25771069
- [Derived] Huang X, Liu L, Song Y, Gao L, Zhao M, Bao H, Qin X, Wu Y, Wu Q, Bi C, Yue A, Fang C, Ma H, Cui Y, Tang G, Li P, Zhang Y, Li J, Wang B, Xu X, Wang H, Parati G, Spence JD, Wang X, Huo Y, Chen G, Cheng X; investigators of intensive BP control in China. Achieving blood pressure control targets in hypertensive patients of rural China - a pilot randomized trial. Trials. 2020 Jun 11;21(1):515. doi: 10.1186/s13063-020-04368-1. PMID 32527283